CLINICAL TRIAL: NCT01341054
Title: Chamomilla Recutita Use of Oral Mucositis in Patients Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Use of Chamomilla Recutita in Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fernanda Titareli Merizio Martins Braga, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: uspchamomilla01
Record Dates: First submitted 2011-04-19; First posted 2011-04-25 (Estimated); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Mucositis
Keywords: mucositis; chamomilla; therapeutics
MeSH Terms: conditions — Mucositis | interventions — Mouthwashes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- mouthwash with Chamomilla extract 1% (Experimental): The Chamomile recutita mouthwash 1% was administered two times daily for 30 days.
  Interventions: Other: mouthwash with Chamomilla
- mouthwash with Chamomilla extract 2% (Experimental): The Chamomile recutita mouthwash 2% was administered two times daily for 30 days.
  Interventions: Other: mouthwash with Chamomilla
- standard oral care protocol (Active Comparator): The standard protocol at the unit, which comprises mouthwash with chlorhexidine 0,12%; oral hygiene teaching. In case the toothbrush cannot be used due to gingival or oral mucosa bleeding, gauze is used to replace it.
  Interventions: Other: Standard oral care protocol
- mouthwash with Chamomilla extract 0.5% (Experimental): The Chamomile recutita mouthwash 0.5% was administered two times daily for 30 days, starting on the first day of chemotherapy.
  Interventions: Other: mouthwash with Chamomilla

INTERVENTIONS:
Other: mouthwash with Chamomilla — The Chamomile recutita mouthwash was administered two times daily for 30 days. 10 mL of this solution was swished around in the mouth for approximately one minute and then expectorated.
  Arms: mouthwash with Chamomilla extract 0.5%; mouthwash with Chamomilla extract 1%; mouthwash with Chamomilla extract 2%
Other: Standard oral care protocol — The standard protocol at the unit, which comprises mouthwash with chlorhexidine 0,12% twice a day; oral hygiene teaching, recommended at least three times per day and always after meals. For brushing, brushes with extra-soft bristles and non-abrasive toothpaste are used. In case the toothbrush cannot be used due to gingival or oral mucosa bleeding, gauze is used to replace it.
  Arms: standard oral care protocol

SUMMARY:
To determine the Chamomilla recutita solution dose needed to reduce the intensity and evolution time of oral mucositis in adult subjects submitted to HSCT.

DETAILED DESCRIPTION:
Population: adult subjects, submitted to hematopoietic stem cell transplantation (HSCT) at a cancer hospital in the interior of São Paulo State. The following inclusion criteria were adopted for sample selection purposes: subjects over 18 years of age, candidates for allogeneic HSCT and with intact oral cavity on the first day of conditioning. Subjects will be excluded if they present any adverse reaction to the active principles of Chamomilla recutita; receive oral or intravenous anticoagulation therapy; use oral or systemic topical anti-inflammatory medication; receive any other type of intervention for mucositis not included in the standard oral care protocol.

ELIGIBILITY:
Inclusion Criteria:

* subjects over 18 years of age;
* candidates for allogeneic HSCT;
* with intact oral cavity on the first day of conditioning.

Exclusion Criteria:

* present any adverse reaction to the active principles of Chamomilla recutita;
* receive oral or intravenous anticoagulation therapy;
* use oral or systemic topical anti-inflammatory medication;
* receive any other type of intervention for mucositis not included in the standard oral care protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Oral mucositis intensity | The measurement will be held on the first day of the conditioning regimen to bone marrow grafting. In an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda TM Braga, RN, Principal Investigator — University of Sao Paulo; Emilia C Carvalho, Study Director — University of Sao Paulo
Locations (1):
- Hospital Amaral Carvalho, Jaú, São Paulo, Brazil

REFERENCES:
- [Background] Braga FT, Santos AC, Bueno PC, Silveira RC, Santos CB, Bastos JK, Carvalho EC. Use of Chamomilla recutita in the Prevention and Treatment of Oral Mucositis in Patients Undergoing Hematopoietic Stem Cell Transplantation: A Randomized, Controlled, Phase II Clinical Trial. Cancer Nurs. 2015 Jul-Aug;38(4):322-9. doi: 10.1097/NCC.0000000000000194. PMID 25232958
- See also: PubMed — https://www.ncbi.nlm.nih.gov/pubmed/25232958